CLINICAL TRIAL: NCT03226977
Title: Nasal Intermittent Positive Pressure Ventilation vs Continuous Positive Airway Pressure for Preterm Infants With Respiratory Distress Syndrome:a Multicenter Randomized Controlled Study
Brief Title: Nasal Intermittent Positive Pressure Ventilation(NIPPV) vs Continuous Positive Airway Pressure for Respiratory Distress Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Collaborators: Guiyang Maternity and Child Health Care Hospital (Other); Children's Hospital of Chongqing Medical University (Other); Chongqing Maternal and Child Health Hospital (Other); Yan'an Affiliated Hospital of Kunming Medical University (Other); The Children's Hospital of Zhejiang University School of Medicine (Other); Chengdu Women's and Children's Central Hospital (Other); Kunming Children's Hospital (Other); Shanxi Provincial Maternity and Children's Hospital (Other); Children's Hospital of Fudan University (Other); Guangdong Women and Children Hospital (Other); Nanjing Children's Hospital (Other); Jiulongpo No.1 People's Hospital (Other)
Responsible Party: Principal Investigator, Ma Juan, Principal Investigator, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NIPPV of multicenter
Record Dates: First submitted 2017-07-12; First posted 2017-07-24 (Actual); Last update posted 2017-07-24 (Actual); Status verified 2017-06

CONDITIONS: Nasal Intermittent Positive Pressure Ventilation; Nasal Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NIPPV (Experimental): NIPPV is used as a primary mode of ventilation in premature infants with respiratory distress syndrome
  Interventions: Device: NIPPV
- NCPAP (Active Comparator): NCPAP is used as a primary mode of ventilation in premature infants with respiratory distress syndrome
  Interventions: Device: NCPAP

INTERVENTIONS:
Device: NIPPV — NIPPV is used as a primary mode of ventilation in premature infants with respiratory distress syndrome
  Arms: NIPPV
Device: NCPAP — NCPAP is used as a primary mode of ventilation in premature infants with respiratory distress syndrome
  Arms: NCPAP

SUMMARY:
In the past, several studies have compared the effects between nasal intermittent positive pressure ventilation(NIPPV) and nasal continuous positive airway pressure(NCPAP) on the incidence of intubation in preterm infants, and the results were inconsistent.The purpose of the present study was to compare NIPPV with NCPAP on the need for endotracheal ventilation and subsequent complications

DETAILED DESCRIPTION:
To this day, early use of noninvasive respiratory support strategies has been suggested to be the most effective pathway to reduce those risks. Nasal continuous positive airway pressure (NCPAP) and nasal intermittent positive pressure ventilation (NIPPV) are two widely used ways of noninvasive ventilation strategies in preterm infant. As compared with invasive ventilation, NCPAP reduces the risks abnormal neurodevelopment. However, there is only 60% success rate of avoiding intubation in the preterm neonate supported with NCPAP. Supplying with an intermittent peak pressure on NCPAP, NIPPV is considered as a strengthened version of NCPAP with increased flow delivery in the upper airway, increased minute volume and functional residual capacity and recruitment of collapsed alveoli, improved stability of the chest wall and reduced asynchrony of thoraco-abdominal movement,which have been proven to be crucial to decrease the incidences of invasive ventilation and death. However, studies have compared the effects between nasal intermittent positive pressure ventilation(NIPPV) and nasal continuous positive airway pressure(NCPAP) on the incidence of intubation in preterm infants, and the results were inconsistent.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age (GA) is from 26 to 37 weeks;
* Diagnosis of RDS. The diagnosis of respiratory distress syndrome(RDS) will be based on clinical manifestations (tachypnea, nasal flaring and or grunting) and chest X-ray findings;
* RDS Silverman score>5;
* Informed parental consent has been obtained.

Exclusion Criteria:

* Severe RDS requiring early intubation according to the American Academy of Pediatrics guidelines for neonatal resuscitation;
* Major congenital malformations or complex congenital heart disease;
* Group B hemolytic streptococcus pneumonia, septicemia, pneumothorax, pulmonary hemorrhage;
* Cardiopulmonary arrest needing prolonged resuscitation;
* Transferred out of the neonatal intensive care unit without treatment.

Ages: 5 Minutes to 6 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1000 (Estimated)
Dates: Start 2017-08-01 (Estimated); Primary Completion 2020-07-30 (Estimated); Study Completion 2020-07-30 (Estimated)

PRIMARY OUTCOMES:
intubation rate | within 7 days
  the infant is intubated ventilation

SECONDARY OUTCOMES:
Intraventricular hemorrhage | within 28 days
  the incidence of intraventricular hemorrhage
bronchopulmonary dysplasia | at a post-menstrual age of 36 weeks or at discharge
  bronchopulmonary dysplasia was defined according to the National Institutes of Health consensus definition
Bayley Scales of Infant Development | at 2 months old and 2 years old
  scores of Bayley Scales of Infant Development
Neonatal necrotizing enterocolitis(NEC) | within 7 days
  the incidence of neonatal necrotizing enterocolitis(>stage II);for NEC, Bell staging will be used

CONTACTS AND LOCATIONS:
Overall Officials: Shi Yuan, PhD,MD, Study Director — Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Locations (1):
- Department of Pediatrics, Daping Hospital, Third Military Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided